CLINICAL TRIAL: NCT00562809
Title: A Multicenter, Open-Label Study Assessing the Efficacy and Safety of Irbesartan 150/12.5 mg and 300/25 mg in Patients With Hypertension Not Controlled by Monotherapy
Brief Title: The Efficacy and Safety of Irbesartan 150/12.5 mg and 300/25 mg in Patients With Mild Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8829
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

INTERVENTIONS:
Drug: IRBESARTAN — 150/12.5 mg tablets one or two tablets orally per day

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Irbesartan 150/12.5 mg and 300/25 mg in patients with hypertension not controlled by monotherapy.

DETAILED DESCRIPTION:
The primary and secondary endpoints applied to sub-groups defined by age, race, diabetes, metabolic syndrome and prior HTN therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have hypertension and uncontrolled SBP on monotherapy.
* Patients who have read, signed and received a copy of the informed consent prior to any study procedures

Note: Female patients must be post-menopausal for one year, surgically sterilized, or using a medically accepted method of contraception (intrauterine device, oral contraceptives, barrier method with spermicide) and must agree to use an effective method of contraception throughout the study.

Exclusion Criteria:

* Any history of secondary hypertension
* History of hypertensive encephalopathy, stroke, or transient ischemic attack (TIA) within the past 12 months
* History of myocardial infarction, percutaneous transluminal coronary revascularization, coronary artery bypass graft, and/or unstable angina pectoris within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2003-07; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Change in the mean SBP | from baseline to week 18

SECONDARY OUTCOMES:
Change in mean DBP | from baseline to week 18.
Changes in mean SBP and DBP | from baseline to week 10
SBP and DBP response and control rates | at weeks 10 and 18

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mooney, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States